CLINICAL TRIAL: NCT03751228
Title: An Open-Label Taste Assessment of BMS-986165 in Healthy Participants
Brief Title: A Taste Assessment of BMS-986165 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-068
Record Dates: First submitted 2018-11-06; First posted 2018-11-23 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Healthy Participants
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986165 taste evaluation (Experimental): BMS-986165 taste evaluation using Active Pharmaceutical Ingredient (API) and Prototypes of the API containing various flavors and sweeteners
  Interventions: Drug: BMS-986165; Drug: Active Pharmaceutical Ingredient

INTERVENTIONS:
Drug: BMS-986165 — Swish and expectorate after tasting
Drug: Active Pharmaceutical Ingredient — Swish and expectorate after tasting
  Other Names: API

SUMMARY:
The purpose of this study is to assess the taste characteristics of BMS-986165 formulations, alone and mixed, in order to develop a pediatric oral form of BMS-986165.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* WOCBP must agree to follow instructions for method(s) of contraception for 5 half-lives of BMS-986165 (2 days) plus 30 days (duration of ovulatory cycle) for a total of 32 days after each tasting day.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception 5 half-lives of the study drug (2 days) after each tasting day.

Exclusion Criteria:

* A known sensitivity to BMS-986165
* A history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the participant. This may include but is not limited to: a history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; or history of mental disease

Other protocol defined inclusion/exclusion criteria could apply

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Taste properties of BMS-986165 alone & in prototypes to determine Aromatic identity will be measured using the Flavor Profile of the Flavor Leadership Criteria | Approximately 2 years
Taste properties of BMS-986165 alone & in prototypes to determine amplitude will be measured using the Flavor Profile of the Flavor Leadership Criteria | Approximately 2 years
Taste properties of BMS-986165 alone & in prototypes to determine mouth-feel will be measured using the Flavor Profile of the Flavor Leadership Criteria | Approximately 2 years
Taste properties of BMS-986165 alone & in prototypes to determine off-notes will be measured using the Flavor Profile of the Flavor Leadership Criteria | Approximately 2 years
Taste properties of BMS-986165 alone & in prototypes to determine aftertaste will be measured using the Flavor Profile of the Flavor Leadership Criteria | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Senopsys, Woburn, Massachusetts, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm